CLINICAL TRIAL: NCT01461057
Title: An Open-Label, Randomized, Multicenter Phase IIa Study Evaluating Pertuzumab in Combination With Trastuzumab and Chemotherapy in Patients With HER2-Positive Advanced Gastric Cancer
Brief Title: A Study of Pertuzumab in Combination With Trastuzumab and Chemotherapy in Patients With HER2-Positive Advanced Gastric Cancer
Acronym: JOSHUA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP27836
Record Dates: First submitted 2011-10-26; First posted 2011-10-27 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Cisplatin; pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pertuzumab 840/420 mg (Experimental): Participants received pertuzumab as an intravenous (IV) infusion at a loading dose of 840 milligrams (mg) for cycle 1 and a dose of 420 mg every three weeks (Q3W) for cycles 2-6. Participants in both arms received trastuzumab, cisplatin, and capecitabine. Capecitabine 1000 milligram per meter squared (mg/m^2) was administered orally twice daily, from the evening of Day 1 to the morning of Day 15 of each cycle. Cisplatin 80 mg/m^2 was administered as an IV infusion on Day 1 of each cycle. Trastuzumab was administered as an IV infusion at a loading dose of 8 mg/kg for Cycle 1 and a dose of 6 milligram per kilogram (mg/kg) Q3W for subsequent cycles.
  Interventions: Drug: Capecitabine; Drug: Cisplatin; Drug: Pertuzumab; Drug: Trastuzumab
- Pertuzumab 840/840 mg (Experimental): Participants received 840 mg as an IV infusion Q3W for cycles 1-6. Participants in both arms received trastuzumab, cisplatin, and capecitabine. Capecitabine 1000 mg/m^2 was administered orally twice daily, from the evening of Day 1 to the morning of Day 15 of each cycle. Cisplatin 80 mg/m^2 was administered as an IV infusion on Day 1 of each cycle. Trastuzumab was administered as an IV infusion at a loading dose of 8 mg/kg for Cycle 1 and a dose of 6 mg/kg Q3W for subsequent cycles.
  Interventions: Drug: Capecitabine; Drug: Cisplatin; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Capecitabine — 1000 mg/m2 twice daily, from the evening of Day 1 to the morning of Day 15 of each cycle
  Other Names: Xeloda
Drug: Cisplatin — 80 mg/m2 on Day 1 of each cycle
Drug: Pertuzumab — loading dose of 840 mg, then 420 mg once every three weeks
  Other Names: Perjeta
  Arms: Pertuzumab 840/420 mg
Drug: Pertuzumab — 840 mg once every three weeks
  Other Names: Perjeta
  Arms: Pertuzumab 840/840 mg
Drug: Trastuzumab — loading dose of 8 mg/kg for Cycle 1 and a dose of 6 mg/kg for subsequent cycles
  Other Names: Herceptin

SUMMARY:
This randomized, multicenter, open-label study will evaluate two different doses of pertuzumab in combination with Herceptin (trastuzumab) and chemotherapy in the first-line treatment of participants with metastatic HER2-positive adenocarcinoma of the stomach or gastroesophageal junction. Participants will be randomized in a 1:1 ratio to two treatment arms. Participants in the Pertuzumab 840/420 mg Arm will receive a pertuzumab loading dose of 840 mg for Cycle 1 and a dose of 420 mg for Cycles 2-6, and participants in the Pertuzumab 840/840 mg Arm will receive pertuzumab 840 mg for all six cycles. Participants in both treatment arms will receive trastuzumab, cisplatin, and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, greater than or equal to (>=) 18 of age
* Adenocarcinoma of the stomach or gastroesophageal junction with inoperable locally advanced or metastatic disease, not amenable to curative therapy
* Measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST), v1.1
* HER2-positive tumor
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 3 months

Exclusion Criteria:

* Previous chemotherapy for advanced or metastatic disease (except (prior adjuvant or neoadjuvant therapy at least 6 months before enrollment in the study)
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Active (significant or uncontrolled) gastrointestinal bleeding
* Abnormal laboratory values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12-06 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Czechia (5):
  - Masaryk Memorial Cancer Institute; Oncological Clinic, Brno
  - Fakultni Nemocnice Hradec Kralove; Dept of Radiotherapy & Oncology, Hradec Králové
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - Fakultní Nemocnice V Motole; Radioterapeuticko-Onkologicke Oddeleni, Prague
  - University Hospital Na Bulovce; Institut of Radiation Oncology, Prague
- France (3):
  - Hopital Morvan, Brest
  - CRLCC Val dAurelle Paul Lam, Montpellier
  - Hopital Robert Debre; DERMATOLOGIE, Reims
- Germany (4):
  - Charité-Universitätsm. Berlin; Med. Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunolo., Berlin
  - Klinikum Braunschweig; Medizinische Klinik III; Klinik für Hämatologie und Onkologie, Braunschweig
  - Krankenhaus Nordwest; Klinik f. Onkologie und Hämatologie, Frankfurt
  - Klinikum Mannheim III. Medizinische Klinik, Mannheim
- Italy (3):
  - Campus Universitario S.Venuta; Centro Oncologico T.Campanella, Catanzaro, Calabria
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - A.O. Universitaria Pisana; Oncologia, Pisa, Tuscany
- Academish Ziekenhuis Maastricht (Azm); Inwendige Geneeskunde, Maastricht, Netherlands
- South Korea (3):
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Yonsei Medical Center; Dept. of Medicine , Division of Hemato-Oncology, Seoul
  - Asan Medical Center; Medical Oncology, Seoul
- Spain (3):
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pertuzumab 840/420 mg | Pertuzumab 840/840 mg
Started | 15 | 15
Completed | 0 | 0
Not Completed | 15 | 15
Not completed — Death | 10 | 9
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Physician Decision | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Progression of Disease | 1 | 0
Not completed — Study Terminated by Sponsor | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pertuzumab 840/420 mg | Pertuzumab 840/840 mg | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Customized [Count of Participants; unit: Participants]
  18 - 40 years | 2 | 1 | 3
  41 - 64 years | 4 | 9 | 13
  Greater than or equal to (>=) 65 years | 9 | 5 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Day 43 Serum Pertuzumab Trough Concentrations (Cmin) Greater Than or Equal to (>=) 20 Microgram Per Milliliter (mcg/mL)
Time Frame: Day 43
Population: The primary pharmacokinetic (PK) analysis population consisted of all participants with a measurable PK samples on Day 43.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab 840/420 mg | Pertuzumab 840/840 mg
Number analyzed (Participants) | 15 | 12
percentage of participants | 91.6 [78.3 to 99.2] | 98.3 [91.4 to 99.97]

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered the investigational product which does not necessarily have a causal relationship with this treatment.
Time Frame: From randomization of first participant to end of study (approximately 6 years)
Population: Safety population included all participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Pertuzumab 840/420 mg | Pertuzumab 840/840 mg
Number analyzed (Participants) | 15 | 15
participants | 15 | 15

ADVERSE EVENTS:
Time Frame: From randomization of first participant to end of study (approximately 6 years)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered the investigational product which does not necessarily have a causal relationship with this treatment.
Arm/Group | Pertuzumab 840/420 mg | Pertuzumab 840/840 mg
All-Cause Mortality (participants affected / at risk) | 10/15 | 9/15
Serious Adverse Events (participants affected / at risk) | 11/15 | 10/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab 840/420 mg (N=15) | Pertuzumab 840/840 mg (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Biliary sepsis (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Myoglobin blood increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Food intolerance (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab 840/420 mg (N=15) | Pertuzumab 840/840 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 9 | 11
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 14 | 11
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 5
Enteritis (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 13
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Stomatits (Gastrointestinal disorders) | 9 | 6
Tooth loss (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 6 | 3
Catheter site pain (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 2
Chills (General disorders) | 2 | 1
Face oedema (General disorders) | 2 | 1
Fatigue (General disorders) | 5 | 7
General physical health deterioration (General disorders) | 0 | 1
Influenza like illness (General disorders) | 2 | 0
Injection site reaction (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 4 | 2
Oedema peripheral (General disorders) | 5 | 4
Pain (General disorders) | 1 | 3
Pyrexia (General disorders) | 6 | 2
Xerosis (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 2
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Herpes Simplex (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1
Oral herpes (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Tinea versicolour (Infections and infestations) | 0 | 1
Toxocariasis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 3
Amylase increased (Investigations) | 0 | 1
Aspartate aminotransferase inreased (Investigations) | 1 | 2
Bilirubin conjugated increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 2
Blood cholesterol increased (Investigations) | 1 | 0
Blood cholinesterase decreased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood fibrinogen increased (Investigations) | 1 | 0
Blood iron increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 4 | 1
Ejection fraction decreased (Investigations) | 2 | 0
Fibrin D dimer increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 11 | 11
Platelet count decreased (Investigations) | 1 | 2
Protein total decreased (Investigations) | 2 | 0
Prothrombin time shortened (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 4 | 4
Weight increased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 11 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 3
Hyposideraemia (Metabolism and nutrition disorders) | 2 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 1 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Ageusia (Nervous system disorders) | 0 | 1
Cholinergic syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 8 | 3
Dysgeusia (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Neurotoxicity (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 4
Polyneuropathy (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Affective disorder (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 4 | 2
Sleep disorder (Psychiatric disorders) | 0 | 1
Somatic symptom disorder (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 3 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 | 3
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Vitamin D decreased (Investigations) | 1 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.